CLINICAL TRIAL: NCT04246333
Title: Feasibility and Safety of Duodenal Feeds in Very Low Birth Weight Infants
Brief Title: Duodenal Feeds in Very Low Birth Weight Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00217658
Record Dates: First submitted 2020-01-22; First posted 2020-01-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: BPD - Bronchopulmonary Dysplasia; VLBW - Very Low Birth Weight Infant; Feeding Disorder Neonatal; Feeding; Difficult, Newborn; Premature Birth; Chronic Lung Disease of Prematurity
Keywords: Duodenal feeds; Transpyloric feeds; Bronchopulmonary Dysplasia; BPD; Premature infant; Neonate
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric Feeds (No Intervention): Patients in this arm will receive feeds via the standard route which is gastric feeds.
- Duodenal Feeds (Experimental): Patients in this arm will receive feeds via the experimental route which is duodenal feeds.
  Interventions: Other: Mode of Delivery of Feeds

INTERVENTIONS:
Other: Mode of Delivery of Feeds — Eligible infants will be recruited and enrolled and randomized to either duodenal feeds (DF) or gastric feeds (GF), which will occur just prior to the infants advancing beyond 50mL/kg/day of enteral feeds. All enrolled infants will be fed per our institutional feeding protocol. Once infants advance past a volume of 50mL/kg/day of enteral feeds, at this point infants will be randomized to DF or GF groups.
  Arms: Duodenal Feeds

SUMMARY:
Premature infants have high rates of bronchopulmonary dysplasia (BPD) due to prematurity of the participants' lungs and the need for prolonged respiratory support. These infants are at increased risk for gastroesophageal reflux and aspiration which may exacerbate lung injury. Transpyloric feeds, specifically duodenal feeds, may be used to bypass the stomach and directly feed the duodenum decreasing the amount of gastric reflux contributing to aspiration. Duodenal feeds are equivalent to gastric feeds with regards to nutritional outcomes, and have been shown to decrease events of apnea and bradycardia in premature infants. This study will evaluate the feasibility and safety of duodenal feeds in premature infants. The hypothesis is that duodenal feeds may be safely and successfully performed in premature very low birth weight infants.

DETAILED DESCRIPTION:
The primary outcome of this study is the safety and feasibility of duodenal feeds in very low birth weight infants. The secondary outcomes are various measures related to growth, respiratory support, comorbidities, and hospitalization.

Eligibility of infants admitted to the Johns Hopkins All Children's Neonatal Intensive Care Unit (NICU) will be determined based on inclusion and exclusion criteria. Eligible infants will be recruited and enrolled by 14 days of life after informed consent is obtained. Randomization of the infants into two groups- investigational continuous Duodenal Feeds (DF) or standard Gastric Feeds (GF) - will occur just prior to the infants advancing beyond 50mL/kg/day of enteral feeds.

All enrolled infants will be fed per the institutional feeding protocol. Once infants advance past 50mL/kg/day of enteral feeds, at this point infants will be randomized to DF or GF groups in a 1:1 block randomization using blinded envelopes. Multiple gestation infants will be randomized individually.

Placement of gastric tubes will be per standard of practice, and insertion of duodenal tube will be per manual of operations. Continuous duodenal feeds will be provided over 24 hours as a continuous infusion through a nasoduodenal or oro-duodenal tube. Standard gastric feeds will be infused via a nasogastric or orogastric tube per the instructions of the medical team. Gastric feeds are provided as standard of care in the NICU; intermittent bolus feeds over 15-60 minutes. Feeding time may be prolonged by the medical team, for longer than 60 minutes and possibly even be given continuously, for various reasons (emesis, reflux, apnea, bradycardia, etc.) and will be monitored and recorded. Feed volume and advancement will continue to be determined by standardized institutional feeding guidelines. Decision to provide further fortification of feeds beyond institutional guidelines will be determined by the medical team and not standardized in this protocol. Once full enteral feeds are achieved (total fluid goal of at least 140mL/kg/day), patients will continue to receive feeds via the designated route.

An institutional "Infant Driven Feeding Guideline" is utilized to evaluate readiness to orally feed and to transition premature infants from enteral to oral feeds. Once an infant is eligible to receive oral feeds per this guideline (32 weeks postmenstrual age, and tolerating ≤2L flow via nasal cannula for at least 24 hours), the study will allow the medical team to transition infants in the DF group to gastric feeds. Regarding transitioning infant from duodenal to gastric feeds, infants are initially placed on continuous gastric feeds, and once the participants have demonstrated tolerance (no evidence of reflux, increased respiratory support, emesis), the participants are then transitioned to bolus gastric feeds progressively. Infants may be allowed to orally feed during this transition period if the participants meet the appropriate infant driven feeding scores per protocol.

All infants in this study will be monitored for primary and secondary outcomes through the duration of admission and up until the time of discharge. Safety events will be frequently monitored for throughout the duration of admission and addressed immediately if warranted.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the Johns Hopkins All Children's NICU before 72 hours of life
* Infants with a birth weight <1251g

Exclusion Criteria:

* First obtained pH <7.0
* APGAR <5 at 5 minutes (The Apgar score is a test given to newborns soon after birth. This test checks a baby's heart rate, muscle tone, and other signs to see if extra medical care or emergency care is needed. Appearance, Pulse, Grimace, Activity, Respiration (APGAR))
* Infants on hydrocortisone for hypotension prior to randomization
* Infants with intrauterine growth restriction (IUGR) defined by birth weight ≤10th percentile for gestational age
* Infants with congenital anomalies, including but not limited to: Chromosomal abnormalities;Structural airway or pulmonary abnormalities (e.g. tracheoesophageal fistulas, cleft palate, congenital pulmonary adenomatous malformation, etc.); Abdominal anomalies requiring surgical interventions (e.g. intestinal atresia, intestinal webs, gastroschisis, omphalocele, anal atresia); Major cardiac anomalies
* Infants with a history of intestinal perforation or NEC
* Presence of gastrostomy tube
* Infants who have not been initiated on any volume of enteral feeds by 10 days of life

Ages: 0 Days to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of successful placements of duodenal tubes | 12 months
  Success to be measured by appropriate placement of the duodenal tube within the duodenum as confirmed by radiographic imaging.
Safety as assessed by number of intestinal perforations | 12 months
  Safety of duodenal feeds in very low birth weight infants as measured by the number of intestinal perforations secondary to placement of duodenal tube.

SECONDARY OUTCOMES:
Supplemental oxygen requirement | duration of hospitalization, up to 15 months
  Number of days on supplemental oxygen >21% throughout duration of hospitalization
Number of participants with Bronchopulmonary Dysplasia | 15 months
  Mild, moderate, severe Bronchopulmonary Dysplasia (BPD) as defined by the NICHD/NHLBI/ORD Workshop published in 2001
Number of deaths during hospitalization | 15 months
Number of days of mechanical ventilation | 15 months
  Days of invasive mechanical ventilation up until hospital discharge
Number of participants with late-onset sepsis | 15 months
  Number of participants diagnosed with Culture-positive sepsis after 72 hours of life
Central line days | 15 months
  Cumulative days of indwelling central venous catheters (peripherally inserted central catheters, tunneled venous catheters, umbilical venous catheters)
Number of participants with necrotizing enterocolitis | 15 months
  Number of participants with necrotizing enterocolitis (NEC) defined by Modified Bells Stage II or greater
Number of replaced enteral tubes | 15 months
  Number of replaced enteral tubes, gastric or duodenal, per patient
Number of Radiographs related to enteral tube placement | 15 months
  Number of radiographs obtained with the indication of enteral tube placement, gastric or duodenal
Weight percentile at 36 weeks postmenstrual age | At 36 weeks
  Weight percentile at 36 weeks postmenstrual age
Height percentile at 36 weeks postmenstrual age | At 36 weeks
  Height percentile at 36 weeks postmenstrual age
Head circumference percentile at 36 weeks postmenstrual age | At 36 weeks
  Head circumference percentile at 36 weeks postmenstrual age
Z-scores for weight at 36 weeks postmenstrual age | At 36 weeks
  Z-scores for weight at 36 weeks postmenstrual age calculated using PediTools
Z-scores for height at 36 weeks postmenstrual age | At 36 weeks
  Z-scores for height at 36 weeks postmenstrual age calculated using PediTools
Z-scores for head circumference at 36 weeks postmenstrual age | At 36 weeks
  Z-scores for head circumference at 36 weeks postmenstrual age calculated using PediTools
Daily daily weight gain | At 36 weeks
  Average daily weight gain (kg/day) calculated from birth until 36 weeks postmenstrual age using the fetal-infant growth reference (FIGR) equation
Length of stay | duration of hospitalization, up to 15 months
  Length of hospital stay (days)
Need for excess fortification of feeds | 15 months
  Number of participants requiring fortification beyond 24kcal/oz
Use of postnatal dexamethasone | 15 months
  Number of participants requiring use of postnatal dexamethasone for respiratory indications
Use of chronic diuretics | 15 months
  Number of participants requiring use of chronic diuretics including thiazide diuretics and spironolactone

CONTACTS AND LOCATIONS:
Overall Officials: Noura Nickel, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Background] Fenton TR, Nasser R, Eliasziw M, Kim JH, Bilan D, Sauve R. Validating the weight gain of preterm infants between the reference growth curve of the fetus and the term infant. BMC Pediatr. 2013 Jun 11;13:92. doi: 10.1186/1471-2431-13-92. PMID 23758808
- [Background] Shennan AT, Dunn MS, Ohlsson A, Lennox K, Hoskins EM. Abnormal pulmonary outcomes in premature infants: prediction from oxygen requirement in the neonatal period. Pediatrics. 1988 Oct;82(4):527-32. PMID 3174313
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] Poets CF. Gastroesophageal reflux: a critical review of its role in preterm infants. Pediatrics. 2004 Feb;113(2):e128-32. doi: 10.1542/peds.113.2.e128. PMID 14754982
- [Background] Omari TI, Barnett CP, Benninga MA, Lontis R, Goodchild L, Haslam RR, Dent J, Davidson GP. Mechanisms of gastro-oesophageal reflux in preterm and term infants with reflux disease. Gut. 2002 Oct;51(4):475-9. doi: 10.1136/gut.51.4.475. PMID 12235066
- [Background] Garland JS, Alex CP, Johnston N, Yan JC, Werlin SL. Association between tracheal pepsin, a reliable marker of gastric aspiration, and head of bed elevation among ventilated neonates. J Neonatal Perinatal Med. 2014 Jan 1;7(3):185-92. doi: 10.3233/NPM-14814020. PMID 25318633
- [Background] Peter CS, Wiechers C, Bohnhorst B, Silny J, Poets CF. Influence of nasogastric tubes on gastroesophageal reflux in preterm infants: a multiple intraluminal impedance study. J Pediatr. 2002 Aug;141(2):277-9. doi: 10.1067/mpd.2002.126298. PMID 12183728
- [Background] Jolley SG, Halpern CT, Sterling CE, Feldman BH. The relationship of respiratory complications from gastroesophageal reflux to prematurity in infants. J Pediatr Surg. 1990 Jul;25(7):755-7. doi: 10.1016/s0022-3468(05)80012-0. PMID 2380892
- [Background] Farhath S, Aghai ZH, Nakhla T, Saslow J, He Z, Soundar S, Mehta DI. Pepsin, a reliable marker of gastric aspiration, is frequently detected in tracheal aspirates from premature ventilated neonates: relationship with feeding and methylxanthine therapy. J Pediatr Gastroenterol Nutr. 2006 Sep;43(3):336-41. doi: 10.1097/01.mpg.0000232015.56155.03. PMID 16954956
- [Background] Knight PR, Davidson BA, Nader ND, Helinski JD, Marschke CJ, Russo TA, Hutson AD, Notter RH, Holm BA. Progressive, severe lung injury secondary to the interaction of insults in gastric aspiration. Exp Lung Res. 2004 Oct-Nov;30(7):535-57. doi: 10.1080/01902140490489162. PMID 15371091
- [Background] Blondheim O, Abbasi S, Fox WW, Bhutani VK. Effect of enteral gavage feeding rate on pulmonary functions of very low birth weight infants. J Pediatr. 1993 May;122(5 Pt 1):751-5. doi: 10.1016/s0022-3476(06)80021-1. PMID 8496756
- [Background] Jensen EA, Munson DA, Zhang H, Blinman TA, Kirpalani H. Anti-gastroesophageal reflux surgery in infants with severe bronchopulmonary dysplasia. Pediatr Pulmonol. 2015 Jun;50(6):584-7. doi: 10.1002/ppul.23052. Epub 2014 Apr 21. PMID 24753497
- [Background] McGuire W, McEwan P. Transpyloric versus gastric tube feeding for preterm infants. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003487. doi: 10.1002/14651858.CD003487.pub2. PMID 17636725
- [Background] Wells DH, Zachman RD. Nasojejunal feedings in low-birth-weight infants. J Pediatr. 1975 Aug;87(2):276-9. doi: 10.1016/s0022-3476(75)80602-0. PMID 807697
- [Background] Drew JH, Johnston R, Finocchiaro C, Taylor PS, Goldberg HJ. A comparison of nasojejunal witn nasogastric feedings in low-birth-weight infants. Aust Paediatr J. 1979 Jun;15(2):98-100. doi: 10.1111/j.1440-1754.1979.tb01198.x. No abstract available. PMID 114157
- [Background] Roy RN, Pollnitz RB, Hamilton JR, Chance GW. Impaired assimilation of nasojejunal feeds in healthy low-birth-weight newborn infants. J Pediatr. 1977 Mar;90(3):431-4. doi: 10.1016/s0022-3476(77)80710-5. PMID 402459
- [Background] Whitfield MF. Poor weight gain of the low birthweight infant fed nasojejunally. Arch Dis Child. 1982 Aug;57(8):597-601. doi: 10.1136/adc.57.8.597. PMID 6810764
- [Background] Sullivan S, Schanler RJ, Kim JH, Patel AL, Trawoger R, Kiechl-Kohlendorfer U, Chan GM, Blanco CL, Abrams S, Cotten CM, Laroia N, Ehrenkranz RA, Dudell G, Cristofalo EA, Meier P, Lee ML, Rechtman DJ, Lucas A. An exclusively human milk-based diet is associated with a lower rate of necrotizing enterocolitis than a diet of human milk and bovine milk-based products. J Pediatr. 2010 Apr;156(4):562-7.e1. doi: 10.1016/j.jpeds.2009.10.040. Epub 2009 Dec 29. PMID 20036378
- [Background] Laing IA, Lang MA, Callaghan O, Hume R. Nasogastric compared with nasoduodenal feeding in low birthweight infants. Arch Dis Child. 1986 Feb;61(2):138-41. doi: 10.1136/adc.61.2.138. PMID 3082297
- [Background] Wallenstein MB, Brooks C, Kline TA, Beck RQ, Yang W, Shaw GM, Stevenson DK. Early transpyloric vs gastric feeding in preterm infants: a retrospective cohort study. J Perinatol. 2019 Jun;39(6):837-841. doi: 10.1038/s41372-019-0372-3. Epub 2019 Apr 9. PMID 30967655
- [Background] Macdonald PD, Skeoch CH, Carse H, Dryburgh F, Alroomi LG, Galea P, Gettinby G. Randomised trial of continuous nasogastric, bolus nasogastric, and transpyloric feeding in infants of birth weight under 1400 g. Arch Dis Child. 1992 Apr;67(4 Spec No):429-31. doi: 10.1136/adc.67.4_spec_no.429. PMID 1586185
- [Background] Pereira GR, Lemons JA. Controlled study of transpyloric and intermittent gavage feeding in the small preterm infant. Pediatrics. 1981 Jan;67(1):68-72. PMID 6787557
- [Background] Caillie MV, Powell GK. Nasoduodenal versus nasogastric feeding in the very low birthweight infant. Pediatrics. 1975 Dec;56(6):1065-72. PMID 812052
- [Background] Malcolm WF, Smith PB, Mears S, Goldberg RN, Cotten CM. Transpyloric tube feeding in very low birthweight infants with suspected gastroesophageal reflux: impact on apnea and bradycardia. J Perinatol. 2009 May;29(5):372-5. doi: 10.1038/jp.2008.234. Epub 2009 Feb 26. PMID 19242488
- [Background] Misra S, Macwan K, Albert V. Transpyloric feeding in gastroesophageal-reflux-associated apnea in premature infants. Acta Paediatr. 2007 Oct;96(10):1426-9. doi: 10.1111/j.1651-2227.2007.00442.x. Epub 2007 Sep 10. PMID 17850402
- [Background] Hsu CW, Sun SF, Lin SL, Kang SP, Chu KA, Lin CH, Huang HH. Duodenal versus gastric feeding in medical intensive care unit patients: a prospective, randomized, clinical study. Crit Care Med. 2009 Jun;37(6):1866-72. doi: 10.1097/CCM.0b013e31819ffcda. PMID 19384225
- [Result] Radford PJ, Stillwell PC, Blue B, Hertel G. Aspiration complicating bronchopulmonary dysplasia. Chest. 1995 Jan;107(1):185-8. doi: 10.1378/chest.107.1.185. PMID 7813274